CLINICAL TRIAL: NCT07059689
Title: High Flow Nasal Cannula vs. Non-Invasive Ventilation in Post-Extubation Pediatric Cardiac Surgery Patients: A Randomized Controlled Trial
Brief Title: High-Flow Nasal Cannula vs. NIV After Extubation in Children Undergoing Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yogi Prawira, Head of Pediatric Emergency and Intensive Care Divison, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-04-0565
Record Dates: First submitted 2025-06-19; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Heart Defects, Congenital; Intensive Care Units, Pediatric; Respiration, Artificial; Extubation
MeSH Terms: conditions — Heart Defects, Congenital; Respiratory Aspiration | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled trial involving two intervention arms. Pediatric patients post-cardiac surgery admitted to the Cardiac Intensive Care Unit (CICU) at Cipto Mangunkusumo National General Hospital will be randomly assigned in a 1:1 ratio to receive either High Flow Nasal Cannula (HFNC) therapy or Non-Invasive Ventilation (NIV) for post-extubation respiratory support. Each participant will receive only one type of intervention throughout the study.
Masking Description: This is an open-label study. Due to the visible and functional differences between High Flow Nasal Cannula (HFNC) and Non-Invasive Ventilation (NIV), masking of participants, care providers, investigators, and outcomes assessors is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Experimental): Participants in this arm will receive High Flow Nasal Cannula (HFNC) therapy using the Airvo™3 Nasal High Flow System immediately following planned extubation after cardiac surgery.
  Interventions: Device: High Flow Nasal Cannula (HFNC)
- Non-Invasive Ventilation (NIV) (Active Comparator): Participants in this arm will receive Non-Invasive Ventilation (NIV) immediately following planned extubation after cardiac surgery, in accordance with institutional protocols.
  Interventions: Device: Non-Invasive Ventilation (NIV)

INTERVENTIONS:
Device: High Flow Nasal Cannula (HFNC) — Participants in this arm will receive High Flow Nasal Cannula therapy using the Airvo™3 Nasal High Flow System immediately after planned extubation following cardiac surgery
  Arms: High Flow Nasal Cannula
Device: Non-Invasive Ventilation (NIV) — Participants in this arm will receive Non-Invasive Ventilation (NIV) immediately after planned extubation following cardiac surgery. NIV will be delivered using standard ICU ventilator settings, with parameters tailored to each patient's clinical condition
  Arms: Non-Invasive Ventilation (NIV)

SUMMARY:
High-Flow Nasal Cannula vs. NIV After Extubation in Children Undergoing Heart Surgery

DETAILED DESCRIPTION:
This study aims to compare the extubation success rate between the use of High Flow Nasal Cannula (HFNC) and Non-Invasive Ventilation (NIV) in pediatric patients post-cardiac surgery at the Cipto Mangunkusumo National General Hospital. Additionally, this study seeks to identify factors influencing extubation failure in high-risk patient populations, compare CICU length of stay, sedation usage and COMFORT scale between patients receiving HFNC and those receiving NIV.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age.
* Post-cardiac surgery patients in the CICU of Cipto Mangunkusumo National General Hospital
* Patients at high risk of extubation failure (e.g., young age, open sternotomy, mechanical ventilation >48 hours).
* Patients who pass the extubation readiness test and spontaneous breathing trial.

Exclusion Criteria:

* Diaphragmatic paralysis.
* Decreased consciousness.
* Neuromuscular disease.
* Pneumothorax without drainage.
* Airway obstruction.
* Patients with a tracheostomy.
* Unplanned extubation.
* Patient received PEEP (Positive End-Expiratory Pressure) >7 prior to extubation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Requiring Reintubation Within 48 - 72 Hours Following Planned Extubation After Cardiac Surgery | 72 hours post-extubation
  Participants who require reintubation due to respiratory failure, clinical deterioration, or complications related to respiratory support will be recorded. This outcome will be compared between the HFNC and NIV groups to assess extubation success.

SECONDARY OUTCOMES:
Length of Stay in the Cardiac Intensive Care Unit (CICU) | 1 month
  The total number of days each participant remains in the CICU will be recorded and compared between the HFNC and NIV groups.
Total Duration of Sedation Post-Extubation | Up to 72 hours post-extubation
  The cumulative duration (in hours) of sedative medication administration following extubation, measured up to 72 hours post-extubation. Duration will be compared between the HFNC and NIV groups.
Total Dosage of Sedation Post-Extubation | Up to 72 hours post-extubation
  The cumulative total dose (in milligrams) of sedative medications administered following extubation, measured up to 72 hours post-extubation. Dosage will be compared between the HFNC and NIV groups.
Change in COMFORT Scale Scores Post-Extubation | Up to 48 hours post-extubation
  The COMFORT Behavioral Scale will be used to assess patient comfort and distress levels at 0, 6, 12, 18, 24, 30, 36, 42, and 48 hours post-extubation. This scale includes multiple behavioral indicators such as alertness, agitation, crying, physical movement, muscle tone, and facial tension.
  Scores range from 6 to 30, where higher scores indicate greater distress and lower scores indicate better comfort/sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Pediatric Emergency and Intensive Care Divison, Principal Investigator — Indonesia University
Locations (1):
- Faculty of Medicine, University of Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuitunen I, Uimonen M. Noninvasive respiratory support preventing reintubation after pediatric cardiac surgery-A systematic review. Paediatr Anaesth. 2024 Mar;34(3):204-211. doi: 10.1111/pan.14808. Epub 2023 Dec 1. PMID 38041510
- [Background] Elmitwalli I, Abdelhady E, Kalsotra S, Gehred A, Tobias JD, Olbrecht VA. Use of high-flow nasal cannula versus other noninvasive ventilation techniques or conventional oxygen therapy for respiratory support following pediatric cardiac surgery: A systematic review and meta-analysis. Paediatr Anaesth. 2024 Jun;34(6):519-531. doi: 10.1111/pan.14866. Epub 2024 Feb 22. PMID 38389199
- [Background] Zhou SJ, Chen XH, Liu YY, Chen Q, Zheng YR, Zhang QL. Comparison of high-flow nasal cannula oxygenation and non-invasive ventilation for postoperative pediatric cardiac surgery: a meta-analysis. BMC Pulm Med. 2024 Feb 21;24(1):92. doi: 10.1186/s12890-024-02901-5. PMID 38383357
- [Background] McQueen M, Rojas J, Sun SC, Tero R, Ives K, Bednarek F, Owens L, Dysart K, Dungan G, Shaffer TH, Miller TL. Safety and Long Term Outcomes with High Flow Nasal Cannula Therapy in Neonatology: A Large Retrospective Cohort Study. J Pulm Respir Med. 2014 Dec;4(6):216. doi: 10.4172/2161-105X.1000216. PMID 26167395
- [Background] Mayfield S, Bogossian F, O'Malley L, Schibler A. High-flow nasal cannula oxygen therapy for infants with bronchiolitis: pilot study. J Paediatr Child Health. 2014 May;50(5):373-8. doi: 10.1111/jpc.12509. Epub 2014 Feb 25. PMID 24612137
- [Background] Doshi P, Whittle JS, Bublewicz M, Kearney J, Ashe T, Graham R, Salazar S, Ellis TW Jr, Maynard D, Dennis R, Tillotson A, Hill M, Granado M, Gordon N, Dunlap C, Spivey S, Miller TL. High-Velocity Nasal Insufflation in the Treatment of Respiratory Failure: A Randomized Clinical Trial. Ann Emerg Med. 2018 Jul;72(1):73-83.e5. doi: 10.1016/j.annemergmed.2017.12.006. Epub 2018 Jan 6. PMID 29310868
- [Background] Demoule A, Chevret S, Carlucci A, Kouatchet A, Jaber S, Meziani F, Schmidt M, Schnell D, Clergue C, Aboab J, Rabbat A, Eon B, Guerin C, Georges H, Zuber B, Dellamonica J, Das V, Cousson J, Perez D, Brochard L, Azoulay E; oVNI Study Group; REVA Network (Research Network in Mechanical Ventilation). Changing use of noninvasive ventilation in critically ill patients: trends over 15 years in francophone countries. Intensive Care Med. 2016 Jan;42(1):82-92. doi: 10.1007/s00134-015-4087-4. Epub 2015 Oct 13. PMID 26464393
- [Background] Chang CJ, Chiang LL, Chen KY, Feng PH, Su CL, Hsu HS. High-Flow Nasal Cannula versus Noninvasive Positive Pressure Ventilation in Patients with Heart Failure after Extubation: An Observational Cohort Study. Can Respir J. 2020 Jul 3;2020:6736475. doi: 10.1155/2020/6736475. eCollection 2020. PMID 32714476
- [Background] Simeonov L, Pechilkov D, Kaneva A, McLellan MC, Jenkins K. Early extubation strategy after congenital heart surgery: 1-year single-centre experience. Cardiol Young. 2022 Mar;32(3):357-363. doi: 10.1017/S1047951121002067. Epub 2021 Jun 7. PMID 34092274
- [Background] Rooney SR, Mastropietro CW, Benneyworth B, Graham EM, Klugman D, Costello J, Ghanayem N, Zhang W, Banerjee M, Gaies M. Influence of Early Extubation Location on Outcomes Following Pediatric Cardiac Surgery. Pediatr Crit Care Med. 2020 Oct;21(10):e915-e921. doi: 10.1097/PCC.0000000000002452. PMID 32639473
- [Background] Miura S, Butt W, Thompson J, Namachivayam SP. Recurrent Extubation Failure Following Neonatal Cardiac Surgery Is Associated with Increased Mortality. Pediatr Cardiol. 2021 Jun;42(5):1149-1156. doi: 10.1007/s00246-021-02593-2. Epub 2021 Apr 17. PMID 33864485
- [Background] Miura S, Jardim PV, Butt W, Namachivayam SP. Extubation Failure and Major Adverse Events Secondary to Extubation Failure Following Neonatal Cardiac Surgery. Pediatr Crit Care Med. 2020 Dec;21(12):e1119-e1125. doi: 10.1097/PCC.0000000000002470. PMID 32804741
- [Background] Murni IK, Djer MM, Yanuarso PB, Putra ST, Advani N, Rachmat J, Perdana A, Sukardi R. Outcome of pediatric cardiac surgery and predictors of major complication in a developing country. Ann Pediatr Cardiol. 2019 Jan-Apr;12(1):38-44. doi: 10.4103/apc.APC_146_17. PMID 30745768

DOCUMENTS (1):
  • Study Protocol (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT07059689/Prot_000.pdf